CLINICAL TRIAL: NCT06629454
Title: Digital Incentive Spirometer for Assessing Incentive Spirometry Adherence
Brief Title: Digital Incentive Spirometry Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ebebfaib
Record Dates: First submitted 2024-09-25; First posted 2024-10-08 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Function; Incentive Spirometry; Patient Adherence; Lung Resection; Thoracic Surgery
Keywords: Incentive spirometer; Patient adherence; Digital incentive spirometer
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single arm proof of concept study of a digital incentive spirometer (Experimental): This single-arm proof-of-concept research study aims to assess the effect of a digital incentive spirometer (IS) device and a companion mobile-based app on incentive spirometry adherence in patients post-surgery. The digital IS utilizes a sensor to measure inspiratory breaths, and these data are transmitted wirelessly to a secure cloud database. The spirometer and app include a patient reminder system, exercise gamification strategies, progress tracking, and additional features designed to promote patient IS use.
  Interventions: Device: Adherence to digital incentive spirometer in the postop period after major chest surgery.

INTERVENTIONS:
Device: Adherence to digital incentive spirometer in the postop period after major chest surgery. — Major chest surgery can lead to respiratory compromise and traditional breathing exercises are not supervised or monitored. The primary objective of this study is to evaluate the effect of a multifeatured digital IS and integrated phone app on patient adherence to incentive spirometry. Together the device and app will include the following functions: an auditory and haptic reminder cue, visual and auditory cues to guide exercise completion, exercise gamification, and data tracking and visualization features.

SUMMARY:
This single-arm proof-of-concept research study aims to assess the effect of a digital incentive spirometer (IS) device and a companion mobile-based app on incentive spirometry adherence in patients post-surgery. The digital IS utilizes a sensor to measure inspiratory breaths, and these data are transmitted wirelessly to a secure cloud database. The spirometer and app include a patient reminder system, exercise gamification strategies, progress tracking, and additional features designed to promote patient IS use.

DETAILED DESCRIPTION:
Incentive spirometry is frequently prescribed as a standard-of-care for patients post-surgery to reduce the risk of developing postoperative pulmonary complications associated with atelectasis. An incentive spirometer (IS) is a mechanical breathing device that assists with pulmonary rehabilitation through improving lung expansion by encouraging deep breathing. While performing incentive spirometry exercises is effective at lowering atelectasis severity, ventilation time, and pulmonary complication rates, patient adherence to performing exercises is very poor. Medical staff, due to time constraints, often cannot supervise all of their patients' entire incentive spirometry regimens (usually every 10-15 min during wakeful hours), contributing to low adherence and incorrect exercise completion. This is compounded by current incentive spirometers lacking a method for accurately collecting patient exercise and adherence data. The present study seeks to evaluate the effect of a digital IS that provides instruction signals and exercise reminders on patients' incentive spirometry adherence.

This single-arm proof-of-concept research study aims to assess the effect of a digital incentive spirometer (IS) device and a companion mobile-based app on incentive spirometry adherence in patients post-surgery. The digital IS utilizes a sensor to measure inspiratory breaths, and these data are transmitted wirelessly to a secure cloud database. The spirometer and app include a patient reminder system, exercise gamification strategies, progress tracking, and additional features designed to promote patient IS use.

The objective of this study is to evaluate the effect of a digital IS that provides gentle auditory and haptic reminders and exercise guidance on patient adherence to incentive spirometry. Secondarily, this study will evaluate metrics relating to lung function to assess post-surgery lung recovery in patients using the digital IS.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, 18 years or older.
4. Undergoes any anatomic lung resection surgery
5. An incentive spirometer is expected to be ordered for the patient as standard-of-care
6. There is no restriction on active medications.

Exclusion Criteria:

There are no exclusions based on economic status, gender, race, or ethnicity. An individual who meets any of the following criteria will be excluded from participation in this study:

1. Vulnerable populations who in the opinion of the investigator are unable to give Informed Consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy.
2. History of prior non-compliance to prescribed therapy or presence or history of significant psychiatric condition (e.g., drug or alcohol addiction, psychosis, schizophrenia), or cognitive issue which would in the opinion of the investigator, make it difficult for the patient to comply with the study procedures or follow the investigators instructions.
3. Populations for whom in the opinion of the investigator, incentive spirometry is deemed inappropriate due to medical condition or otherwise.
4. Pregnant individuals due to low likelihood of meeting inclusion criteria 4. Licensed medical professionals on the clinical team will follow proper procedures in determining if the individual is consenting. Proper procedures entail doing all of the following: giving a patient adequate information concerning the study, providing adequate opportunity for the patient to consider all options, responding to the patient's questions, ensuring that the patient has comprehended this information, obtaining the patient's voluntary agreement to participate and, continuing to provide information as the patient or situation requires. There will be ample opportunity for the patient to ask questions. In the event that the patient is in a vulnerable population and unable to provide consent, they will not be eligible to participate in the study and thus will not be screened. If the individual is not able to provide informed consent or if consent is not certain due to impairments or other factors, they will not be considered for study participation. In the event that the patient is in a vulnerable population and unable to provide consent, they will not be eligible to participate in the study and thus will not be screened.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-12-27 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doraid Jarrar, MD, Principal Investigator — University of Pennsylvania
Locations (6):
- United States (6):
  - Penn Medicine Cherry Hill, Cherry Hill, New Jersey
  - Penn Medicine Valley Forge, Berwyn, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Medicine University City, Philadelphia, Pennsylvania
  - Penn Thoracic Surgery Presbyterian, Philadelphia, Pennsylvania
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 31 patients enrolled. 30 patients completed per protocol.
Pre-assignment Details: One participant was withdrawn from the study by clinician decision.
Period: Overall Study
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Started | 31
Completed | 30
Not Completed | 1
Not completed — Withdraw by Clinician Decision | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis includes age, sex, height, weight, race, and ethnicity.
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 66 [33 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 22
  More than one race | 0
  Unknown or Not Reported | 1
Height [Mean (Full Range); unit: inches] — Height, weight, and sex is used to calculate a baseline incentive spirometry volume (mL) goal
  inches | 66.7 [62 to 74]
Weight [Mean (Full Range); unit: pounds (lbs)] | 177 [75 to 269]
Procedure Target Lobe [Count of Participants; unit: Participants]
  Right Upper Lobe | 10
  Right Lower Lobe | 8
  Left Upper Lobe | 5
  Left Lower Lobe | 3
  Right Middle Lobe | 1
  More than one lobe | 3
Preoperative Incentive Spirometry Volume [Mean (Full Range); unit: milliliters]
  Average preoperative volume | 2066 [532 to 3941]
  Maximum preoperative volume | 2339 [915 to 4204]
Preoperative Incentive Spirometry Flow Rate [Mean (Full Range); unit: milliliters per second]
  Average flow rate | 259 [161 to 461]
  Maximum flow rate | 386 [235 to 615]

OUTCOME MEASURES:

1. Primary Outcome: Incentive Spirometry Adherence (Breath Attempts Per Day)
Description: Number of inspiratory breath attempts performed with the digital IS per day.
Time Frame: Till discharge or up to 7 days
Measure: Mean (Inter-Quartile Range); unit: Breath attempts
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 30
Breath attempts | 45 [23 to 59]

2. Primary Outcome: Incentive Spirometry Consistency (Hours Per Day With ≥1 Breath)
Description: Number of hours in which at least one inspiratory breath was attempted using the digital IS per day.
Time Frame: Till discharge or up to 7 days
Measure: Mean (Inter-Quartile Range); unit: Hours
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 30
Hours | 7.6 [5.75 to 10]

3. Secondary Outcome: Volume of Inspiratory Breaths Attempted With the Digital IS
Description: Inspiratory volume in milliliters measured from one inhalation from the device
Time Frame: Till discharge or up to 7 days
Measure: Mean (Full Range); unit: milliliters
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 30
milliliters
  Average postoperative volume | 1314 [403 to 2517]
  Maximum postoperative volume | 2375 [716 to 7506]

4. Secondary Outcome: Blood Oxygen Saturation
Description: Average postoperative SpO2 per patient. Mean is the mean across the patient cohort.
Time Frame: Till discharge or up to 7 days
Measure: Mean (Full Range); unit: percentage of oxygen saturation
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 30
percentage of oxygen saturation | 96 [93 to 98]

5. Secondary Outcome: Pain Scores
Description: Postoperative pain scores will be reported on a scale from 0 (no pain) to 10 (unbearable pain). These are then averaged per patient. Mean and range is reported for the entirely of the patient cohort.
Time Frame: Till discharge or up to 7 days
Measure: Mean (Full Range); unit: units on a scale from 0 to 10
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 30
units on a scale from 0 to 10 | 4 [0 to 7]

6. Secondary Outcome: Flow Rate of Inspiratory Breaths Attempted From the Digital IS
Description: Flow rate over time (mL/sec) of each inspiratory breath measured from one inhalation from the device.
Time Frame: Till discharge or up to 7 days
Measure: Mean (Full Range); unit: Milliliters per second
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 30
Milliliters per second
  Average flow rate | 186 [132 to 288]
  Maximum flow rate | 357 [172 to 405]

7. Other Pre Specified Outcome: Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO)
Description: Preoperative diffusing capacity of the lung for carbon monoxide to move from air sacs into the bloodstream as a percent of predicted value based on the person's age, sex, height, and other factors.
Time Frame: up to 2 weeks before the surgery
Measure: Mean (Full Range); unit: percentage of predicted value
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 26
percentage of predicted value | 79.0 [26.1 to 124]

8. Other Pre Specified Outcome: Forced Expiratory Volume in 1 Second (FEV-1)
Description: Preoperative forced expiration volume in 1 second as a percentage of predicted value based on the person's age, sex, height, and other factors.
Time Frame: up to 2 weeks before the surgery
Measure: Mean (Full Range); unit: percentage of predicted value
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 30
percentage of predicted value | 90.6 [21.5 to 129.3]

9. Other Pre Specified Outcome: Forced Vital Capacity (FVC)
Description: Preoperative forced vital capacity of the lungs as a percentage of predicted value based on the person's age, sex, height, and other factors.
Time Frame: up to 2 weeks before the surgery
Measure: Mean (Full Range); unit: percentage of predicted value
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 30
percentage of predicted value | 94.4 [66.3 to 135.5]

10. Other Pre Specified Outcome: Vital Capacity (VC)
Description: Preoperative vital capacity of the lungs.
Time Frame: up to 2 weeks before the surgery
Population: This metric was not collected as part of standard of care pulmonary function testing.
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Residual Volume (RV)
Description: Preoperative residual volume of the lungs as a percentage of predicted value based on the person's age, sex, height, and other factors.
Time Frame: up to 2 weeks before the surgery
Measure: Mean (Full Range); unit: percentage of predicted value
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 20
percentage of predicted value | 108 [75.3 to 203.6]

12. Other Pre Specified Outcome: Total Lung Capacity (TLC)
Description: Preoperative total lung capacity as a percentage of predicted value based on the person's age, sex, height, and other factors.
Time Frame: up to 2 weeks before the surgery
Measure: Mean (Full Range); unit: percentage of predicted value
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 25
percentage of predicted value | 94.1 [74.3 to 123.0]

13. Other Pre Specified Outcome: Forced Expiratory Flow (FEF25-75)
Description: Forced expiratory flow rate between 25% and 75% of the forced vital capacity, pre-bronchodilator, as a percentage of predicted value based on the person's age, sex, height, and other factors.
Time Frame: up to 2 weeks before the surgery
Measure: Mean (Full Range); unit: percentage of predicted value
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 23
percentage of predicted value | 93.9 [8.2 to 189.3]

14. Other Pre Specified Outcome: Thoracic Gas Volume (TGV)
Description: Total gas volume within the chest cavity when the airway is temporarily blocked as a percent of predicted value based on the person's age, sex, height, and other factors.
Time Frame: up to 2 weeks before the surgery
Measure: Mean (Full Range); unit: percentage of predicted value
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 12
percentage of predicted value | 99.9 [74.7 to 155]

15. Other Pre Specified Outcome: Expiratory Reserve Volume (ERV)
Description: Expiratory reserve volume of the lungs as a percentage of predicted value based on the person's age, sex, height, and other factors.
Time Frame: up to 2 weeks before the surgery
Measure: Mean (Full Range); unit: percentage of predicted value
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 14
percentage of predicted value | 95.5 [29.8 to 166.9]

16. Other Pre Specified Outcome: Discharge Survey Responses - Device Engagement
Description: Device engagement survey responses. Patients are instructed on the paper survey to "Circle how much you agree or disagree with the following statements:"
Time Frame: On the day of patient discharge from the hospital, an average of 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 24
Participants
  It was easy to know when to do my exercises with my device.: Strongly Agree | 14
  It was easy to know when to do my exercises with my device.: Agree | 6
  It was easy to know when to do my exercises with my device.: Neutral | 1
  It was easy to know when to do my exercises with my device.: Disagree | 1
  It was easy to know when to do my exercises with my device.: Strongly Disagree | 0
  It was easy to know when to do my exercises with my device.: Incomplete | 2
  It was easy to know when to do my exercises with my device.: Not applicable | 0
  I felt motivated to do my exercises.: Strongly Agree | 7
  I felt motivated to do my exercises.: Agree | 10
  I felt motivated to do my exercises.: Neutral | 5
  I felt motivated to do my exercises.: Disagree | 0
  I felt motivated to do my exercises.: Strongly Disagree | 0
  I felt motivated to do my exercises.: Incomplete | 2
  I felt motivated to do my exercises.: Not applicable | 0
  It was easy to click the button on my device to start an exercise when I wanted to.: Strongly Agree | 14
  It was easy to click the button on my device to start an exercise when I wanted to.: Agree | 10
  It was easy to click the button on my device to start an exercise when I wanted to.: Neutral | 0
  It was easy to click the button on my device to start an exercise when I wanted to.: Disagree | 0
  It was easy to click the button on my device to start an exercise when I wanted to.: Strongly Disagree | 0
  It was easy to click the button on my device to start an exercise when I wanted to.: Incomplete | 0
  It was easy to click the button on my device to start an exercise when I wanted to.: Not applicable | 0
  I liked how the device gave spoken (audio) instructions for the exercises.: Strongly Agree | 9
  I liked how the device gave spoken (audio) instructions for the exercises.: Agree | 8
  I liked how the device gave spoken (audio) instructions for the exercises.: Neutral | 3
  I liked how the device gave spoken (audio) instructions for the exercises.: Disagree | 2
  I liked how the device gave spoken (audio) instructions for the exercises.: Strongly Disagree | 1
  I liked how the device gave spoken (audio) instructions for the exercises.: Incomplete | 1
  I liked how the device gave spoken (audio) instructions for the exercises.: Not applicable | 0
  I liked how my nurse/doctor could see my breathing exercise measurements.: Strongly Agree | 11
  I liked how my nurse/doctor could see my breathing exercise measurements.: Agree | 8
  I liked how my nurse/doctor could see my breathing exercise measurements.: Neutral | 2
  I liked how my nurse/doctor could see my breathing exercise measurements.: Disagree | 0
  I liked how my nurse/doctor could see my breathing exercise measurements.: Strongly Disagree | 1
  I liked how my nurse/doctor could see my breathing exercise measurements.: Incomplete | 2
  I liked how my nurse/doctor could see my breathing exercise measurements.: Not applicable | 0
  I was able to set up the app easily.: Strongly Agree | 6
  I was able to set up the app easily.: Agree | 5
  I was able to set up the app easily.: Neutral | 0
  I was able to set up the app easily.: Disagree | 0
  I was able to set up the app easily.: Strongly Disagree | 0
  I was able to set up the app easily.: Incomplete | 2
  I was able to set up the app easily.: Not applicable | 11
  I liked the app features.: Strongly Agree | 3
  I liked the app features.: Agree | 6
  I liked the app features.: Neutral | 3
  I liked the app features.: Disagree | 0
  I liked the app features.: Strongly Disagree | 0
  I liked the app features.: Incomplete | 2
  I liked the app features.: Not applicable | 10

17. Other Pre Specified Outcome: Discharge Survey Responses - Previous Incentive Spirometry
Description: Have you used an incentive spirometer prior to this hospital stay?
Time Frame: On the day of patient discharge from the hospital, an average of 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 24
Participants
  YES | 7
  NO | 12
  Incomplete | 5

18. Other Pre Specified Outcome: Discharge Survey Responses - Exercise Completion Self-Reported Adherence
Description: Discharge Survey Question: How much of you exercises do you think you completed?
Time Frame: On the day of patient discharge from the hospital, an average of 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
Number analyzed (Participants) | 24
Participants
  0-20%, Close to none | 0
  21-40%, A few of them | 2
  41-60%, Around half | 7
  61-80%, More than half | 9
  81-100%, Almost all | 6
  Incomplete | 0

ADVERSE EVENTS:
Time Frame: From Enrollment Until 4 Months After Discharge, up to 18 weeks
Arm/Group | Single Arm Proof of Concept Study of a Digital Incentive Spirometer
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
This was a single-arm, open-label study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT06629454/Prot_SAP_000.pdf
  • Informed Consent Form (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT06629454/ICF_001.pdf